CLINICAL TRIAL: NCT07156955
Title: Proprioceptive Error Correction Technique Development to Promote Post-stroke Upper Limbs Motor Rehabilitation
Brief Title: Proprioceptive Error Correction for Post-Stroke Upper Limb Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sungkyunkwan University (Other)
Responsible Party: Principal Investigator, Hangue Park, Associate professor, Sungkyunkwan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-06-075-001
Record Dates: First submitted 2025-08-11; First posted 2025-09-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Proprioception
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Electrical stimulation cue first (Experimental): Patients undergo three types of interventions, following one of two processes. Each process has its own protocol in the following order Electrical stimulation cue, Visual cue, and No cue or Electrical stimulation cue, No cue, and Visual cue.
  Interventions: Behavioral: Electrical stimulation cue; Behavioral: Visual stimulation cue; Behavioral: No cue
- Visual stimulation cue first (Experimental): Patients undergo three types of interventions, following one of two processes. Each process has its own protocol in the following order: Visual cue, Electrical stimulation cue, and No cue, or Visual cue, No cue, and Electrical stimulation cue.
  Interventions: Behavioral: Electrical stimulation cue; Behavioral: Visual stimulation cue; Behavioral: No cue
- No cue first (Experimental): Patients undergo three types of interventions, following one of two processes. Each process has its own protocol in the following order: No cue, Electrical stimulation cue, and Visual cue, or No cue, Visual cue, and Electrical stimulation cue.
  Interventions: Behavioral: Electrical stimulation cue; Behavioral: Visual stimulation cue; Behavioral: No cue
- Only electrical stimulation cue (Experimental): Patients undergo one types of interventions which is the Electrical stimulation cue.
  Interventions: Behavioral: Electrical stimulation cue
- Only visual stimulation cue (Experimental): Patients undergo one types of interventions which is the Visual stimulation cue.
  Interventions: Behavioral: No cue
- Only no cue (Experimental): Patients undergo one types of interventions which is the No cue.
  Interventions: Behavioral: Visual stimulation cue

INTERVENTIONS:
Behavioral: Electrical stimulation cue — A single 30-minute session is provided. Electrodes are attached to the cubital fossa, and stimulation is delivered at a frequency that increases up to 70 Hz as the elbow joint approaches the target angle. Target angles are set between 0 degrees and 120 degrees, based on each participant's available range of motion determined during the initial assessment. Participants adjust their elbow joint angle to match the provided target angle using feedback from the electrical stimulation. When the elbow joint angle matches the target angle, the maximum frequency is applied to the cubital fossa. Participants match their elbow joint angle to the target angle based on the given frequency.
  Arms: Electrical stimulation cue first; No cue first; Only electrical stimulation cue; Visual stimulation cue first
Behavioral: Visual stimulation cue — A single 30-minute session is provided. The difference between the current elbow joint angle and the pre-set target angle is displayed on a screen using two colored needles (a red needle for the target angle and a black needle for the current elbow joint angle). The target angle is set within each participant's available range of motion based on the initial assessment. Participants continue the intervention by adjusting their elbow angle using the visual feedback. When the elbow joint angle matches the target angle, the two needles overlap. Based on this visual cue, participants adjust their elbow joint angle to match the target angle.
  Arms: Electrical stimulation cue first; No cue first; Only no cue; Visual stimulation cue first
Behavioral: No cue — A single 30-minute session is provided. The target angle is determined within each participant's available range of motion based on the initial assessment. Throughout the session, participants receive verbal feedback from the assessor and adjust their elbow joint angle accordingly to match the target angle.
  Arms: Electrical stimulation cue first; No cue first; Only visual stimulation cue; Visual stimulation cue first

SUMMARY:
The investigators aim to develop sensory transformation and augmentation technologies that minimize the impact of proprioceptive errors, thereby significantly enhancing motor learning and rehabilitation of the upper limbs. This study is designed to test proprioceptive error compensation techniques in stroke patients.

The human nervous system often receives mismatched information from vision and proprioception during upper limb control, resulting in conflicting sensory inputs that limit the effectiveness of motor learning. In other words, real-time sensory feedback - a critical component of motor learning in the nervous system - is not reliably delivered. Therefore, this study seeks to resolve sensory conflicts by providing additional sensory information through electrical stimulation, with the goal of dramatically improving the effectiveness of motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic or hemorrhagic stroke
* Stroke confirmed by CT or MRI
* Stroke patients with proprioceptive sensory deficits
* Chronic stroke patients with onset at least 3 months prior
* Able to voluntarily flex and extend the elbow joint
* Age 19 years or older
* Provide written informed consent (participant or legal representative)

Exclusion Criteria:

* Severe pain during elbow joint movement
* Elbow joint contracture, spasticity, ataxia, musculoskeletal disorders, fractures, - non-healing ulcers, or open wounds
* Progressive or unstable stroke
* Presence of unilateral neglect
* Coexisting severe neurological disorders
* Major psychiatric disorders such as major depressive disorder, schizophrenia, bipolar disorder, or dementia Presence of a pacemaker

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in upper limb motor function | 6 visits over 3 weeks
  Upper limb motor function will be evaluated using standardized clinical scales such as the Fugl-Meyer Assessment and proprioceptive accuracy tests.
  0 indicates severe movement limitation, while a score of 66 reflects normal motor function of upper limb.
  Participants will undergo evaluations and treatment during six visits over approximately three weeks.

SECONDARY OUTCOMES:
Proprioceptive accuracy | Baseline before intervention and immediately after the 30-minute training session
  Assessment of improvements in upper limb motor function and proprioceptive accuracy after applying sensory error correction techniques in stroke patients. Motor performance will be evaluated using standardized clinical scales and joint position sense tests. The expected outcome measures are a reduction of the error angle relative to the target angle to within ±5 degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Shinchon Severance Rehabilitation Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT07156955/Prot_000.pdf